CLINICAL TRIAL: NCT01378117
Title: Randomized Controlled Study of Dipeptidyl Peptidase-4 (DPP4) Inhibitor (Sitagliptin) Therapy in the Inpatient Management of Patients With Type 2 Diabetes
Brief Title: Dipeptidyl Peptidase-4 Inhibitor (Sitagliptin) Therapy in the Inpatients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Guillermo Umpierrez, MD, Professor of Medicine, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00048954a; NCT01373268 (obsolete NCT alias)
Record Dates: First submitted 2011-03-07; First posted 2011-06-22 (Estimated); Results first posted 2014-06-12 (Estimated); Last update posted 2018-12-07 (Actual); Status verified 2018-11

CONDITIONS: Type 2 Diabetes Mellitus; Hospitalization; Hyperglycemia
Keywords: diabetes; non critical care setting; hyperglycemia; treatment; oral antidiabetic agents; subcutaneous insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Diabetes Mellitus | interventions — Sitagliptin Phosphate; Insulin Glargine; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sitagliptin + SSI prn (Experimental): Sitagliptin once daily plus supplemental doses of lispro if needed using sliding scale insulin (SSI). 100 mg/day (at any time of day) for patients with GFR 50-100 ml/min and 50 mg/day for patients with GFR 30-50 ml/min
  Interventions: Drug: Sitagliptin
- Sitagliptin and glargine+ SSI (Experimental): Sitagliptin 50-100 mg per oral once a day and SubCutaneous (SQ) glargine insulin once daily + correctional doses of lispro if needed for elevated blood glucose using sliding scale insulin (SSI). 100 mg/day (at any time of day) for patients with glomerular filtration rate (GFR) 50-100 ml/min and 50 mg/day for patients with GFR 30-50 ml/min
  Interventions: Drug: glargine
- Glargine and Lispro + SSI (Active Comparator): Glargine once daily and lispro before meals supplemental insulin lispro as needed for elevated blood glucose using sliding scale insulin (SSI)
  Interventions: Drug: lispro

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 50-100mg po once daily
  Other Names: Januvia
  Arms: Sitagliptin + SSI prn
Drug: glargine — glargine once daily
  Other Names: Lantus (glargine)
  Arms: Sitagliptin and glargine+ SSI
Drug: lispro — lispro before meals
  Other Names: Humalog (lispro)
  Arms: Glargine and Lispro + SSI

SUMMARY:
The study is a multicenter, prospective, open-label, randomized pilot study to investigate the safety and efficacy of sitagliptin (Januvia) for the inpatient management of type 2 diabetes (T2D) in general medicine and surgery patients.

DETAILED DESCRIPTION:
High blood glucose levels in hospitalized patients with diabetes are associated with increased risk of medical complications and death. Improved glucose control with insulin injections may improve clinical outcome and prevent some of the hospital complications. Glargine (Lantus®) insulin injection is the most common treatment of diabetes in the hospital. Sitagliptin (Januvia®)is effective in lowering blood glucose, but has not been tested in the hospital. It is not known if sitagliptin is as effective in controlling blood sugars in the hospital. This study will compare sitagliptin by mouth, insulin (glargine) injection, and the combination of sitagliptin and lantus insulin in controlling blood sugar in hospitalized patients with diabetes.

In this pilot study, patients with known history of diabetes treated with diet and/or oral anti-diabetics or with low total daily dose insulin therapy (<0.4 unit/kg/day) will be randomized to receive sitagliptin once daily (group 1), sitagliptin plus basal (glargine) insulin once daily (group 2), or basal bolus regimen with glargine once daily and lispro insulin before meals (group 3). If needed, patients in the 3 treatment groups will receive correction doses of rapid-acting lispro (Humalog®) insulin in the presence of hyperglycemia (BG > 140 mg/dl) per sliding scale. The overall hypothesis is that treatment with sitagliptin once daily alone or in combination with basal insulin in patients with type 2 diabetes will result in a similar improvement in glycemic control and in a lower frequency of hypoglycemic events than treatment with basal bolus insulin regimen with glargine once daily and lispro insulin before meals.

A total of 90 subjects with type 2 diabetes will be recruited in this study. Patients will be recruited at Grady Memorial Hospital and Emory University Hospital.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between the ages of 18 and 80 years admitted to a general medicine and surgery services.
2. A known history of type 2 diabetes mellitus > 3 months, receiving either diet alone, oral antidiabetic agents: sulfonylureas and metformin as monotherapy or in combination therapy (excluding Trazodone (TZDs) and DPP4 inhibitors), or low-dose (≤ 0.4 units/kg/day) insulin therapy.
3. Subjects with a BG >140 mg and < 400 mg/dL without laboratory evidence of diabetic ketoacidosis (serum bicarbonate < 18 milliequivalent /L or positive serum or urinary ketones).

Exclusion Criteria:

1. Age < 18 or > 80 years.
2. Subjects with increased blood glucose concentration, but without a known history of diabetes (stress hyperglycemia).
3. Subjects with a history of type 1 diabetes (suggested by BMI < 25 requiring insulin therapy or with a history of diabetic ketoacidosis and hyperosmolar hyperglycemic state, or ketonuria) [46].
4. History of TZD treatment (pioglitazone or rosiglitazone) or DPP4 inhibitor (sitagliptin or saxagliptin) during the past 3 months prior to admission.
5. Acute critical illness or coronary artery bypass graft (CABG) surgery expected to require prolonged admission to a critical care unit (ICU, cardiac care unit , surgical intensive care unit, neuro ICU).
6. Subjects with gastrointestinal obstruction or adynamic ileus or those expected to require gastrointestinal suction.
7. Medical or surgical patients expected to be kept nil per os (NPO) for >24-48 hours after admission or after completion of surgical procedure.
8. Patients with clinically relevant pancreatic or gallbladder disease.
9. Patients with congestive heart failure (NYHA class III and IV), acute myocardial infarction, clinically significant hepatic disease or significantly impaired renal function (serum creatinine ≥ 2.0 mg/dL).
10. Treatment with oral or injectable corticosteroid.
11. Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
12. Female subjects are pregnant or breast feeding at time of enrollment into the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University SOM
Locations (2):
- United States (2):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

REFERENCES:
- [Result] Umpierrez GE, Gianchandani R, Smiley D, Jacobs S, Wesorick DH, Newton C, Farrokhi F, Peng L, Reyes D, Lathkar-Pradhan S, Pasquel F. Safety and efficacy of sitagliptin therapy for the inpatient management of general medicine and surgery patients with type 2 diabetes: a pilot, randomized, controlled study. Diabetes Care. 2013 Nov;36(11):3430-5. doi: 10.2337/dc13-0277. Epub 2013 Jul 22. PMID 23877988

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 90 patients admitted to general medicine and surgery services in 2012 were enrolled in this pilot study. This study was conducted at Grady Memorial Hospital (Atlanta, GA), Emory University Hospital, and University of Michigan Health System.
Pre-assignment Details: Patients were included if they had Type 2 Diabetes with a BG 140-400 mg/dL and were treated at home with diet, oral antidiabetics, or low-dose insulin. 8 patients were excluded from further analysis because they received <24 h of insulin treatment, were transferred to the ICU, or received corticosteroid therapy.
Groups:
- Sitagliptin + SSI Prn: Sitagliptin once daily plus supplemental doses of lispro if needed.
- Sitagliptin and Glargine+ SSI: Sitagliptin 50-100 mg po once a day and Subcutaneous glargine insulin once daily + correctional doses of lispro if needed for elevated blood glucose using sliding scale Insulin (SSI)
- Glargine and Lispro + SSI: Glargine once daily and lispro before meals + supplemental insulin lispro as needed for elevated blood glucose using sliding scale Insulin (SSI)
Period: Overall Study
Arm/Group | Sitagliptin + SSI Prn | Sitagliptin and Glargine+ SSI | Glargine and Lispro + SSI
Started | 31 | 30 | 29
Completed | 27 | 29 | 26
Not Completed | 4 | 1 | 3
Not completed — withdrawal | 2 | 1 | 2
Not completed — discharged before med given | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Sitagliptin and Glargine + SSI: Sitagliptin 50-100 mg po once a day and subcutaneous glargine insulin once daily + correctional doses of lispro if needed for elevated blood glucose using sliding scale Insulin (SSI)
- Total: Total of all reporting groups
Arm/Group | Sitagliptin + SSI Prn | Sitagliptin and Glargine + SSI | Glargine and Lispro + SSI | Total
Number analyzed (Participants) | 27 | 29 | 26 | 82
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 22 | 23 | 22 | 67
  >=65 years | 5 | 6 | 4 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (11) | 58 (12) | 57 (10) | 58 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 16 | 8 | 34
  Male | 17 | 13 | 18 | 48
Region of Enrollment [Number; unit: participants]
  United States | 27 | 29 | 26 | 82

OUTCOME MEASURES:

1. Primary Outcome: Mean Blood Glucose Levels Among the Three Groups at the Time of Hospitalization to 1st Day After Therapy
Description: The primary outcome of the study is to determine differences in glycemic control as measured by mean BG concentration between sitagliptin once daily and basal bolus therapy with glargine once daily plus supplemental lispro insulin in hospitalized patients with type 2 diabetes mellitus, at the time of admission to the blood glucose levels 24hrs after the therapy
Time Frame: Admission and after 1st day of therapy
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Sitagliptin + SSI Prn | Sitagliptin and Glargine + SSI | Glargine and Lispro + SSI
Number analyzed (Participants) | 27 | 29 | 26
mg/dl
  At time of admission | 209 (67) | 203 (48) | 225 (74)
  After 1st day of therapy | 168.4 (35) | 154.2 (29) | 158.3 (31)

2. Secondary Outcome: Number of Patients With Hypoglycemic Events Among the Treatment Groups
Description: Hypoglycemia is defined as blood glucose (BG) reading <70 mg/dl. The number of hypoglycemia events during hospitalization are recorded and compared among the different groups. BG was measured before each meal and at bedtime (or every 6 h if a patient was not eating) using a point-of-care glucose meter
Time Frame: during hospitalization,up to 10 days
Measure: Count of Participants; unit: Participants
Groups:
- Sitagliptin and Glargine + SSI: Sitagliptin 50-100 mg po once a day and subcutaneous (SQ) glargine insulin once daily + correctional doses of lispro if needed for elevated blood glucose using sliding scale Insulin (SSI)
  glargine: glargine once daily
Arm/Group | Sitagliptin + SSI Prn | Sitagliptin and Glargine + SSI | Glargine and Lispro + SSI
Number analyzed (Participants) | 27 | 29 | 26
Participants | 1 | 2 | 2

3. Secondary Outcome: Number of Patients With Severe Hypoglycemic Episodes Among the 3 Treatment Groups
Description: severe hypoglycemic episodes are defined as blood glucose levels <40 mg/dl. The number of patients with these events during the 5 days of hospitalization are recorded and compared. BG was measured before each meal and at bedtime (or every 6 h if a patient was not eating) using a point-of-care glucose meter.
Time Frame: during hospitalization,up to 5 days
Measure: Count of Participants; unit: Participants
Groups:
- Sitagliptin and Glargine + SSI: Sitagliptin 50-100 mg po once a day and SQ glargine insulin once daily + correctional doses of lispro if needed for elevated blood glucose using sliding scale Insulin (SSI)
Arm/Group | Sitagliptin + SSI Prn | Sitagliptin and Glargine + SSI | Glargine and Lispro + SSI
Number analyzed (Participants) | 27 | 29 | 26
Participants | 0 | 0 | 0

4. Secondary Outcome: Number of Patients With a Mean Daily BG > 240 mg/dL After the 1st Day of Treatment Among the Treatment Groups
Description: Mean daily blood glucose levels are measured to assess the treatment Failures. For study purpose Treatment failure was defined as having three or more consecutive Blood Glucose (BG) readings > 240 mg/dL or a mean daily BG >240 mg/dL after the 1st day of treatment. Number of patients with a mean daily BG > 240 mg/dL after the 1st day of treatment are recorded and compared among the treatment groups. BG was measured before each meal and at bedtime (or every 6 h if a patient was not eating) using a point-of-care glucose meter.
Time Frame: during hospitalization,up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin + SSI Prn | Sitagliptin and Glargine + SSI | Glargine and Lispro + SSI
Number analyzed (Participants) | 27 | 29 | 26
Participants | 3 | 1 | 2

5. Secondary Outcome: Mean Total Daily Dose of Insulin in Units/Day Given During Hospitalization Among the Three Groups
Description: The total insulin includes total glargine insulin (units/day) and total lispro insulin (units/day) given to subjects for maintaining blood glucose levels during hospitalization in different groups. The goal of therapy was to maintain a fasting and premeal glucose concentration between 100 and 140 mg/dL. The doses of insulin were adjusted daily according to protocol. The mean amount is calculated among the different groups and compared.
Time Frame: during hospitalization, up to 10 days
Measure: Mean (Standard Deviation); unit: units/day
Arm/Group | Sitagliptin + SSI Prn | Sitagliptin and Glargine + SSI | Glargine and Lispro + SSI
Number analyzed (Participants) | 27 | 29 | 26
units/day | 11.5 (7) | 28.2 (12) | 39.8 (22)

6. Secondary Outcome: Mean Length of Stay in Days in the Hospital Among Different Groups
Description: The duration of stay in days in the hospital between the three groups is calculated and mean number of days is measured.
Time Frame: during hospitalization, up to 10 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sitagliptin + SSI Prn | Sitagliptin and Glargine + SSI | Glargine and Lispro + SSI
Number analyzed (Participants) | 27 | 29 | 26
days | 6.3 (3) | 6.9 (3) | 6.3 (3)

7. Secondary Outcome: Number of Subjects With Acute Renal Failure Among the Three Randomized Groups During Hospitalization
Description: Acute renal failure is defined as a clinical diagnosis of acute renal failure with documented new-onset abnormal renal function (serum creatinine > 2.2 mg/dL or an increment > 0.5 mg/dL from baseline). The total daily dose of insulin and sitagliptin will be adjusted as per serum creatinine concentration. The total daily insulin dose will be reduced to 0.3 unit/kg in patients with creatinine >1.7 mg/dl. The dose of sitagliptin will be reduced to 50 mg/day in patients with creatinine clearance between 30-50 ml/min (approximate serum creatinine levels >1.7 and ≤3.0 mg/dl for men and >1.5 and ≤2.5 mg/dl for women).
Time Frame: during hospitalization, up to 10 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin + SSI Prn | Sitagliptin and Glargine + SSI | Glargine and Lispro + SSI
Number analyzed (Participants) | 27 | 29 | 26
Participants | 0 | 0 | 0

8. Secondary Outcome: Number of Deaths Among the Subjects in Different Groups
Description: Mortality is defined as death occurring during admission among the participants. The number of deaths in each assigned group is calculated.
Time Frame: during hospitalization, up to 10 days
Measure: Count of Participants; unit: Participants
Groups:
- Glargine and Lispro + SSI: Glargine once daily and lispro before meals + supplemental insulin lispro as needed for elevated blo0d glucose using sliding scale Insulin (SSI)
Arm/Group | Sitagliptin + SSI Prn | Sitagliptin and Glargine + SSI | Glargine and Lispro + SSI
Number analyzed (Participants) | 27 | 29 | 26
Participants | 0 | 0 | 0

9. Secondary Outcome: Percent of Blood Glucose Readings Within Target Range Between 70 and 140 mg/dL Among the Three Groups After 24 Hrs of Randomized Treatment
Description: The blood glucose within target range is defined as the levels between 70 mg/dL and 140 mg/dL. BG was measured before each meal and at bedtime (or every 6 h if a patient was not eating) using a point-of-care glucose meter (ACCUCHECK; Roche, Indianapolis, IN). In addition, BG was measured at any time if a patient experienced symptoms of hypoglycemia or if requested by the treating physician. the percentage of the readings are calculated and compared
Time Frame: during hospitalization, up to 10 days
Measure: Mean (Standard Deviation); unit: percentage of blood glucose readings
Arm/Group | Sitagliptin + SSI Prn | Sitagliptin and Glargine + SSI | Glargine and Lispro + SSI
Number analyzed (Participants) | 27 | 29 | 26
percentage of blood glucose readings | 36 (30) | 43 (28) | 43 (26)

ADVERSE EVENTS:
Time Frame: The time frame includes the number of days the subjects stayed in the hospital, the maximum was up to 10 days.
Description: Please note that 8 patients did not receive study medication because they either withdrew or were discharged prior to receiving study medication; thus the number of participants at risk is 90-8=82 (as stated).
Arm/Group | Sitagliptin + SSI Prn | Sitagliptin and Glargine + SSI | Glargine and Lispro + SSI
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/29 | 0/26
Serious Adverse Events (participants affected / at risk) | 1/27 | 0/29 | 0/26
Other Adverse Events (participants affected / at risk) | 8/27 | 7/29 | 8/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin + SSI Prn (N=27) | Sitagliptin and Glargine + SSI (N=29) | Glargine and Lispro + SSI (N=26)
Angioedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin + SSI Prn (N=27) | Sitagliptin and Glargine + SSI (N=29) | Glargine and Lispro + SSI (N=26)
Hypoglycemia (Endocrine disorders) | 1 | 2 | 2 — Low blood sugar (hypoglycemia) defined as blood glucose less than 70 mg/dl can occur in 10-30% (10 to 30 patients out of one hundred) in hospital patients treated with insulin.
Hyperglycemia (Endocrine disorders) | 3 | 1 | 2 — Persistent Hyperglycemia high blood glucose levels greater than 240 mg/dl
Pressure Ulcer/Skin Ulcer (General disorders) | 3 (3) | 1 (1) | 1 (1)
Urinary Tract infection (Renal and urinary disorders) | 1 (1) | 2 (2) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 1 (1)
Wound infection (General disorders) | 1 (1) | 0 (0) | 0 (0)
Systematic Infection (General disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study recruited a relatively small number of patients and excluded a large number of patients, which included those admitted to the ICU. Study was not powered to determine differences in hospital complications across the three groups

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No